CLINICAL TRIAL: NCT00652028
Title: A Phase II, Open-Label, Multicenter, Escalating Dose, Study to Determine Pharmacokinetic and Pharmacodynamic Profile of Dexmedetomidine in Pediatric Subjects Ages ≥ 2 Through < 17 Years Old
Brief Title: Pharmacokinetics and Pharmacodynamics of Dexmedetomidine in Pediatrics Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEX-08-01
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2015-08

CONDITIONS: Intubated and Mechanically Ventilated Pediatric Subjects
Keywords: Pharmacokinetics; Pharmacodynamics; Escalating dose; Dexmedotimidine; Intubated; Mechanically ventilated; Pediatrics
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Other): Dose level 1
  Interventions: Drug: Dexmedetomidine, midazolam; fentanyl
- Group 2 (Other): Dose level 2
  Interventions: Drug: Dexmedetomidine, midazolam; fentanyl
- Group 3 (Other): Dose level 3
  Interventions: Drug: Dexmedetomidine, midazolam; fentanyl
- Group 4 (Other): Dose level 4
  Interventions: Drug: Dexmedetomidine, midazolam; fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine, midazolam; fentanyl — Dexmedetomidine for sedation; midazolam for rescue sedation according to label; fentanyl for rescue pain according to the label

SUMMARY:
The objective of this study is to characterize the pharmacokinetic and pharmacodynamic profile of dexmedetomidine administered as an intravenous loading dose followed by a continuous intravenous infusion in pediatric subjects ages ≥2 through <17 years old.

DETAILED DESCRIPTION:
This is a phase II, open-label, multicenter, escalating dose study evaluating the pharmacokinetics and pharmacodynamics of dexmedetomidine in pediatric subjects. The study population consists of initially intubated and mechanically ventilated pediatric subjects, ages ≥2 through <17 years old, that require sedation in an intensive care setting for a minimum of 6 hours. Subjects will be divided into two groups based on age: Group I will consist of subjects ages ≥2 through <6 years old and Group II subjects age ≥6 through <17 years old. Within each group there will be four escalating dosing levels. Both groups can enroll simultaneously; however within each group, the next dose level cannot begin to enroll until all subjects have completed the previous dose level and the Data Safety Monitoring Board (DSMB) has approved enrollment to the next level. The level of sedation will be assessed using the Ramsay Sedation Scale (RSS). Based on these scores, and clinical judgment, additional sedation with midazolam will be administered according to the label. Pain will be assessed using the Faces, Legs, Arms, Cry & Consolability (FLACC) scale. Venous blood samples for pharmacokinetic analysis will be obtained at designated times. The pharmacodynamic and safety measures that will be monitored and the pharmacodynamic impact of dexmedetomidine on tracheal extubation will also be explored if subject is extubated within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Initially intubated and mechanically ventilated pediatric subjects in an intensive care setting anticipated to require a minimum of 6 hours of continuous intravenous sedation.
* Age: subjects must fit into one of the following age ranges at screening:

  * ≥2 years old through <6 years old
  * ≥6 years old through <17 years old
* If female, subject is non-lactating and is either:

  1. Not of childbearing potential, defined as pre-menarche, or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy.
  2. Of childbearing potential but is not pregnant at time of baseline.
* Subject's parent(s) or legal guardian(s) has/have voluntarily signed and dated the informed consent document approved by the Institutional Review Board. Assent will be obtained where age-appropriate and according to state regulations.

Exclusion Criteria:

* Pediatric subjects with neurological conditions that prohibit an evaluation of sedation

  * Diminished consciousness from increased intracranial pressure.
  * Extensive brain surgery (surgery requiring intracranial pressure monitor).
  * Diminished cognitive function per PI's discretion.
  * Subjects with immobility from neuromuscular disease or continuous infusion of neuromuscular blocking agents.
* Weight <10 kg.
* Subjects with second degree or third degree heart block unless subject has a pacemaker or pacing wires.
* Hepatic impairment Serum glutamic pyruvic transaminase/Alanine aminotransferase (SGPT/ALT) >100 U/L
* Hypotension based on repeat assessments prior to starting study drug:

  * Age ≥2 years old through ≤12 years old: systolic blood pressure (SBP) <80 mmHg
  * Age >12 years old through <17 years old: SBP <90 mmHg
* Pre-existing bradycardia prior to starting study drug defined as:

  * Age ≥2 years old through ≤6 years old: ≤70 beats per minute (bpm)
  * Age >6 years old through ≤12 years old: ≤60 bpm
  * Age >12 years old through ≤16 years old: ≤50 bpm
* Acute thermal burns involving more than 15 percent total body surface area.
* Subjects who have a known allergy to dexmedetomidine, midazolam (MDZ) or fentanyl.
* Subjects with a life expectancy that is <72 hours.
* Subjects that are expected to have hemodialysis (continuous hemofiltration) or peritoneal dialysis within 48 hours.
* Subjects who have been treated with α-2 agonists/antagonists within two weeks.
* Subjects with a spinal cord injury above T5.
* Subjects who have received another investigational drug within the past 30 days.
* Subjects on nicotine replacement therapy.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of this clinical study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Miami Children's Hospital, Miami, Florida
  - University of Louisville/Kosair Children's Hospital, Louisville, Kentucky
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- Unidad Cirugia Cardiovascular de Guatemala, Guatemala City, Guatemala

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Dexmedetomidine: Loading dose (IV) 0.25 mcg/kg/hour for 10 minutes; Continuous dose (IV infusion) 0.2 mcg/kg/hour for 6-24 hours
- Dose Level 2: Dexmedetomidine: Loading dose (IV) 0.5 mcg/kg/hour for 10 minutes; Continuous dose (IV infusion) 0.4 mcg/kg/hour for 6-24 hours
- Dose Level 3: Dexmedetomidine: Loading dose (IV) 1.0 mcg/kg/hour for 10 minutes; Continuous dose (IV infusion) 0.7 mcg/kg/hour for 6-24 hours
- Dose Level 4: Dexmedetomidine: Loading dose (IV) 1.0 mcg/kg/hour for 10 minutes; Continuous dose (IV infusion) 2.0 mcg/kg/hour for 6-24 hours
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 16 | 14 | 15 | 14
Completed | 15 | 13 | 14 | 14
Not Completed | 1 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — No Longer Meets Entry Criteria | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Participants who received any amount of study drug were included in the Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Total
Number analyzed (Participants) | 16 | 14 | 15 | 14 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.358 (3.4673) | 7.457 (4.5990) | 8.379 (4.4962) | 7.462 (4.2259) | 7.395 (4.1571)
Age, Customized [Number; unit: participants]
  ≥2 through <6 years | 8 | 6 | 6 | 6 | 26
  ≥6 through <17 years | 8 | 8 | 9 | 8 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 9 | 5 | 32
  Male | 6 | 6 | 6 | 9 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 12 | 12 | 13 | 10 | 47
  More than one race | 2 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC0-t)
Description: Area under the concentration-time curve from time zero to the time of the last measurable concentration (AUC0-t) for Dexmedetomidine
Time Frame: ≤30 min prior to start of loading dose (LD); 5 min before finishing LD; 0.5,1,2 & 4-6 hrs after start of maintenance infusion (MI); 30 min prior to end of MI (within 24 hrs of start of MI); 10 min after end of MI and 0.5,1,2,4 & 10 hrs after end of MI.
Population: Full Evaluable Population: Participants who received study drug infusion for at least 5 hours and had available PK data were included in the full evaluable population. This was the primary population for pharmacokinetic (PK) and pharmacodynamic (PD) analyses.
Measure: Mean (Standard Deviation); unit: picograms*hr/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 14 | 13 | 14 | 14
picograms*hr/mL | 2681.332 (2353.3418) | 6460.576 (3766.4657) | 16992.540 (29927.3911) | 28531.864 (17496.3985)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time Infinity (AUC0-∞)
Description: Area under the concentration-time curve from time zero to the time infinity (AUC0-∞) for Dexmedetomidine
Time Frame: ≤30 min prior to start of the loading dose (LD); 5 min before finishing the LD; 0.5,1,2&4 to 6 hrs after start of maintenance infusion (MI); 30 min prior to end of MI (24 hrs of start of MI); 10 min after end of MI and 0.5,1,2,4&10 hrs after end of MI.
Population: Full Evaluable Population: Participants who received study drug infusion for at least 5 hours and had available PK data were included in the full evaluable population. This was the primary population for PK and PD analyses.
Measure: Mean (Standard Deviation); unit: picograms*hr/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 12 | 13 | 14 | 14
picograms*hr/mL | 3153.518 (3343.3451) | 6673.163 (3781.2183) | 17300.539 (29935.7647) | 28970.541 (17936.8970)

3. Primary Outcome: Observed Peak Plasma Concentration
Description: Observed peak plasma concentration (Cmax) for Dexmedetomidine
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 14 | 13 | 14 | 14
picograms per milliliter | 480.437 (625.9946) | 847.691 (633.7352) | 3385.569 (7384.0699) | 3090.939 (1625.5241)

4. Primary Outcome: Terminal Elimination Half-life (t1/2)
Description: Terminal elimination half-life (t1/2) for Dexmedetomidine
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 12 | 13 | 14 | 14
hour | 1.546 (0.3401) | 1.743 (0.3018) | 2.045 (0.6582) | 2.145 (0.6763)

5. Primary Outcome: Plasma Concentration at Steady State (Css)
Description: Plasma concentration at steady state (Css) for Dexmedetomidine
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 12 | 13 | 14 | 14
picograms per milliliter | 402.026 (535.1718) | 539.848 (166.7423) | 1347.284 (1308.0988) | 2827.144 (1169.4226)

6. Primary Outcome: Volume of Steady State Distribution (Vss)
Description: Volume of steady state distribution (Vss) for Dexmedetomidine
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 12 | 13 | 14 | 14
Litre | 56.808 (44.5127) | 35.246 (25.0233) | 32.789 (22.5478) | 43.652 (30.6577)

7. Primary Outcome: Clearance (CL)
Description: Clearance (CL) for Dexmedetomidine
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre/hour
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 12 | 13 | 14 | 14
Litre/hour | 32.208 (40.3982) | 20.268 (10.3508) | 18.565 (8.6995) | 22.199 (14.1623)

8. Primary Outcome: Level of Sedation Based on Average Ramsay Sedation Scale (RSS) Score
Description: RSS Score range from 1 to 6:
  1. Patient is anxious and agitated or restless, or both.
  2. Patient is cooperative, orientated and tranquil.
  3. Patient responds to command only.
  4. Patient exhibits brisk response to light glabellar (between the eyebrows) tap or loud auditory stimulus.
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus.
  6. Patient exhibits no response to stimulus.
Time Frame: Prior to loading (Baseline), 5 and 10 min during the load, at start of maintenance infusion and every 15 min for 1 hour, hourly during the maintenance period, before and within 5 min after midazolam or fentanyl dose during the dexmedetomidine infusion.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 15 | 13 | 14 | 14
units on a scale | 2.4 (0.96) | 2.8 (0.74) | 2.4 (0.5) | 4.0 (1.04)

9. Primary Outcome: Number of Subjects Who Received Rescue Medication for Sedation (Midazolam) and Analgesics (Fentanyl)
Description: Number of subjects who received rescue medication for Sedation (Midazolam) and analgesics (Fentanyl) while intubated during Treatment Period
Time Frame: During the treatment period (Approximately 24 hours)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 16 | 13 | 14 | 14
participants
  Midazolam | 7 | 7 | 5 | 3
  Fentanyl | 12 | 10 | 13 | 8

ADVERSE EVENTS:
Time Frame: From the start of study drug administration until 24 hours following discontinuation of study drug
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/14 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 11/16 | 12/14 | 10/15 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=16) | Dose Level 2 (N=14) | Dose Level 3 (N=15) | Dose Level 4 (N=14)
Convulsion (Nervous system disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=16) | Dose Level 2 (N=14) | Dose Level 3 (N=15) | Dose Level 4 (N=14)
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 2 | 1
Nodal rhythm (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4 | 2 | 2
Chills (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 4 | 4 | 2 | 3
Serratia infection (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Cardiac enzymes increased (Investigations) | 0 | 0 | 1 | 0
Central venous pressure decreased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Analgesia (Nervous system disorders) | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 3
Withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder distension (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 3 | 3
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No